CLINICAL TRIAL: NCT04853836
Title: Olfactory Disfunction After COVID-19: Conventional Therapy Versus Intervention Treatment With Co-ultraPEALut
Brief Title: Olfactory Disfunction and Co-ultraPEALut
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Of Perugia (Other)
Collaborators: Azienda Ospedaliera Ospedali Riuniti Marche Nord, Italy (Unknown); Federico II University (Other); Humanitas Hospital, Italy (Other); San Giovanni Addolorata Hospital (Other); Policlinico Universitario, Catania (Other); Azienda Ospedaliero-Universitaria Careggi (Other); Azienda Ospedaliero Universitaria di Sassari (Other); Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other); Ospedale Universitario di Genova, Italy (Unknown); Istituto per la Sicurezza Sociale (ISS) della Repubblica di San Marino (Unknown); Ospedale Bufalini di Cesena, Italy (Unknown)
Responsible Party: Principal Investigator, Arianna Di Stadio, Adjunct Professor, University Of Perugia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20112020PGFN
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Anosmia; Covid19; Hyposmia; Parosmia; Treatment Compliance
MeSH Terms: conditions — Anosmia; COVID-19; Olfaction Disorders; Patient Compliance | interventions — co-ultraPEALut

STUDY DESIGN:
Intervention Model Description: Single-blinded randomized clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investor will assign patients to one of the groups before Sniff test evaluation at T0
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Rehabilitation therapy only (control group) (Placebo Comparator): Olfactory training / stimulation through Sniffin' Sticks, administered twice every day (10 minutes session)
  Interventions: Procedure: Olfactory Rehab
- Rehabilitation and treatment with PEA-LUT (Active Comparator): Olfactory training / stimulation through Sniffin' Sticks, plus daily treatment with PEA/Luteolin oral supplement
  Interventions: Combination Product: co-ultraPEALut
- Treatment with PEA-LUT one sachet daily (Active Comparator): Patients in this group only used a single dose of PEA-LUT
  Interventions: Drug: PEA-LUT 1 sachet
- Treatment with PEA-LUT two sachet daily (Active Comparator): Patients in this group only used two doses of PEA-LUT
  Interventions: Drug: PEA-LUT 2 sachet day

INTERVENTIONS:
Combination Product: co-ultraPEALut — Olfactory rehab 10 minutes twice a day for all the observation period + co-ultraPEALut (700 PEA + 70 Luteolin) 1 dose daily.
  Arms: Rehabilitation and treatment with PEA-LUT
Procedure: Olfactory Rehab — Olfactory Rehabilitation10 minutes twice a day for all the observation period
  Arms: Rehabilitation therapy only (control group)
Drug: PEA-LUT 1 sachet — Only 1 sachet day of PEA-LUT no olfactory training
  Arms: Treatment with PEA-LUT one sachet daily
Drug: PEA-LUT 2 sachet day — 2 sachets day of PEA-LUT no olfactory training
  Arms: Treatment with PEA-LUT two sachet daily

SUMMARY:
Olfactory dysfunction is common among patients with Corona-Virus-Infection-Disease (COVID)-19, and up to 30% of patients may report persistent disorders of smell or taste as a long-term sequelae. This randomized-controlled study has addressed to compare the efficacy of neuro-protective and anti-inflammatory agents palmitoylethanolamide (PEA) and Luteolin(Treatment) with control (olfactory training) in a cohort of patients who present persistent smell disorders after resolution from Covid-19 and negative swab for 4 months at least.

DETAILED DESCRIPTION:
Patients ages 18 to 70 years with confirmed history of COVID-19 (positive nasopharyngeal swab for SARS-CoV-2) and subjective olfactory dysfunction persisting ≥ 90 days after follow-up negative COVID-19 nasopharyngeal swab are eligible.

All patients will undergo nasal endoscopic examination to look for presence of polyps, masses, anatomic blockage, or other pathology which presence will require exclusion from the study. Patients then will be evaluated at the baseline with Sniffin' Sticks (Burghardt®, Wedel, Germany) prior to initiating olfactory training and/or supplement treatment (T0). One group received daily olfactory training, patients in the supplement group additionally received a daily oral tablet that contained PEA 700 mg and Luteolin 70 mg (Glialia ®, Epitech pharmaceutical, Milano, Italy), or 1 dose of PEA-LUT only or aTwo Dose of PEA-LUT.

Assessment of olfactory function will be repeated at 30 days, 60 and 90 and 120 days

ELIGIBILITY:
Inclusion Criteria:

* 18 to 90 years with confirmed history of COVID-19 (positive nasopharyngeal swab for SARS-CoV-2)
* subjective olfactory dysfunction persisting ≥ 90 days after follow-up negative COVID-19 nasopharyngeal swab

Exclusion Criteria:

* previous history of olfactory-gustatory disorders
* impaired cognitive function
* history of neurodegenerative disease
* medical therapy with possible effects on olfactory function
* presence of rhinological disorders (sinusitis, rhinosinusitis, sinonasal polyposis, atrophic rhinitis, allergy)
* history of chemo-radiotherapy of the head and neck region
* history of stroke or neurotrauma
* severe nasal blockage from stenosis of deformity
* severe psychiatric illness (e.g. schizophrenia, bipolar disorder, olfactory hallucination)
* previous sinonasal
* nasopharyngeal tumors.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Recovery of smell | T1 (30 days), T2 (60 days), T3 (90 days)
  Change of Sniff scores from T0.The Sniffin' Sticks battery was administered following a previously established protocol, using pen-like devices filled with odorants.Three score subtests were conducted to measure olfactory function:
  1. detection threshold ("T", the lowest concentration at which an odor can be perceived),
  2. odor discrimination ("D", ability to distinguish between odors) and
  3. odor identification ("I" ability to assign names to odors). Possible scores ranged from 1-16 for the detection threshold subtest and 0-16 for both the discrimination and identification subtests. Adding these for yielded a TDI "Sniff score." Anosmia was defined as a score of <17, hyposmia by a score 17 to 30.75, and normosmia by a score of ≥31

SECONDARY OUTCOMES:
Parosmia after treatment | 60 days (T2) and 90 days (T3)
  Prevalence of anosmia among the groups in the recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Multicentric, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
Shared, only anonymized data directly requested to PI
Supporting Information: Study Protocol, SAP
Access Criteria: request to PI

REFERENCES:
- [Background] Ralli M, Di Stadio A, Greco A, de Vincentiis M, Polimeni A. Defining the burden of olfactory dysfunction in COVID-19 patients. Eur Rev Med Pharmacol Sci. 2020 Apr;24(7):3440-3441. doi: 10.26355/eurrev_202004_20797. No abstract available. PMID 32329813
- [Background] Meinhardt J, Radke J, Dittmayer C, Franz J, Thomas C, Mothes R, Laue M, Schneider J, Brunink S, Greuel S, Lehmann M, Hassan O, Aschman T, Schumann E, Chua RL, Conrad C, Eils R, Stenzel W, Windgassen M, Rossler L, Goebel HH, Gelderblom HR, Martin H, Nitsche A, Schulz-Schaeffer WJ, Hakroush S, Winkler MS, Tampe B, Scheibe F, Kortvelyessy P, Reinhold D, Siegmund B, Kuhl AA, Elezkurtaj S, Horst D, Oesterhelweg L, Tsokos M, Ingold-Heppner B, Stadelmann C, Drosten C, Corman VM, Radbruch H, Heppner FL. Olfactory transmucosal SARS-CoV-2 invasion as a port of central nervous system entry in individuals with COVID-19. Nat Neurosci. 2021 Feb;24(2):168-175. doi: 10.1038/s41593-020-00758-5. Epub 2020 Nov 30. PMID 33257876
- [Background] Levy JM. Treatment Recommendations for Persistent Smell and Taste Dysfunction Following COVID-19-The Coming Deluge. JAMA Otolaryngol Head Neck Surg. 2020 Aug 1;146(8):733. doi: 10.1001/jamaoto.2020.1378. No abstract available. PMID 32614399
- [Background] D'Ascanio L, Pandolfini M, Cingolani C, Latini G, Gradoni P, Capalbo M, Frausini G, Maranzano M, Brenner MJ, Di Stadio A. Olfactory Dysfunction in COVID-19 Patients: Prevalence and Prognosis for Recovering Sense of Smell. Otolaryngol Head Neck Surg. 2021 Jan;164(1):82-86. doi: 10.1177/0194599820943530. Epub 2020 Jul 14. PMID 32662745
- [Background] Chiu A, Fischbein N, Wintermark M, Zaharchuk G, Yun PT, Zeineh M. COVID-19-induced anosmia associated with olfactory bulb atrophy. Neuroradiology. 2021 Jan;63(1):147-148. doi: 10.1007/s00234-020-02554-1. Epub 2020 Sep 15. PMID 32930820
- [Background] Laurendon T, Radulesco T, Mugnier J, Gerault M, Chagnaud C, El Ahmadi AA, Varoquaux A. Bilateral transient olfactory bulb edema during COVID-19-related anosmia. Neurology. 2020 Aug 4;95(5):224-225. doi: 10.1212/WNL.0000000000009850. Epub 2020 May 22. No abstract available. PMID 32444492
- [Background] Lee MH, Perl DP, Nair G, Li W, Maric D, Murray H, Dodd SJ, Koretsky AP, Watts JA, Cheung V, Masliah E, Horkayne-Szakaly I, Jones R, Stram MN, Moncur J, Hefti M, Folkerth RD, Nath A. Microvascular Injury in the Brains of Patients with Covid-19. N Engl J Med. 2021 Feb 4;384(5):481-483. doi: 10.1056/NEJMc2033369. Epub 2020 Dec 30. No abstract available. PMID 33378608
- [Background] Stoyanov GS, Petkova L, Dzhenkov DL, Sapundzhiev NR, Todorov I. Gross and Histopathology of COVID-19 With First Histology Report of Olfactory Bulb Changes. Cureus. 2020 Dec 4;12(12):e11912. doi: 10.7759/cureus.11912. PMID 33415060
- [Background] Skaper SD, Facci L, Giusti P. Glia and mast cells as targets for palmitoylethanolamide, an anti-inflammatory and neuroprotective lipid mediator. Mol Neurobiol. 2013 Oct;48(2):340-52. doi: 10.1007/s12035-013-8487-6. Epub 2013 Jun 28. PMID 23813098
- [Background] Paniz-Mondolfi A, Bryce C, Grimes Z, Gordon RE, Reidy J, Lednicky J, Sordillo EM, Fowkes M. Central nervous system involvement by severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2). J Med Virol. 2020 Jul;92(7):699-702. doi: 10.1002/jmv.25915. PMID 32314810
- [Background] Guida F, Luongo L, Boccella S, Giordano ME, Romano R, Bellini G, Manzo I, Furiano A, Rizzo A, Imperatore R, Iannotti FA, D'Aniello E, Piscitelli F, Sca Rossi F, Cristino L, Di Marzo V, de Novellis V, Maione S. Palmitoylethanolamide induces microglia changes associated with increased migration and phagocytic activity: involvement of the CB2 receptor. Sci Rep. 2017 Mar 23;7(1):375. doi: 10.1038/s41598-017-00342-1. PMID 28336953
- [Background] Tan D, Yu X, Chen M, Chen J, Xu J. Lutein protects against severe traumatic brain injury through anti-inflammation and antioxidative effects via ICAM-1/Nrf-2. Mol Med Rep. 2017 Oct;16(4):4235-4240. doi: 10.3892/mmr.2017.7040. Epub 2017 Jul 20. PMID 28731190
- [Derived] O'Byrne L, Webster KE, MacKeith S, Philpott C, Hopkins C, Burton MJ. Interventions for the treatment of persistent post-COVID-19 olfactory dysfunction. Cochrane Database Syst Rev. 2022 Sep 5;9(9):CD013876. doi: 10.1002/14651858.CD013876.pub3. PMID 36062970